CLINICAL TRIAL: NCT05686603
Title: Comparison of 1064nm Nd:YAG Picosecond Lasers Using Fractional Micro-lens Array vs. Ablative Fractional 2940nm Er:YAG Lasers for the Treatment of Atrophic Acne Scar in Asians: a 20-week Prospective, Randomized, Split-face, Controlled Trial
Brief Title: Comparison of Picosecond Lasers vs. Ablative Fractional Er:YAG Lasers in Treating Atrophic Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20220419
Record Dates: First submitted 2023-01-09; First posted 2023-01-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-04

CONDITIONS: Acne; Atrophic Scar
Keywords: atrophic scar; acne; picosecond laser; ablative laser; efficacy; safety
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: This prospective, randomized, split-face, controlled trial. Enrolled participant was randomized to receive split-face treatment with fractional 1064-nm Nd:YAG picosecond lasers (PicocareTM, Wontech, Korea) on one side and ablative fractional 2940-nm Er:YAG laser (Dermablate MCL31, Asclepion Laser Technologies, Germany) on the other side. The block randomization was used to assign the treatment modality.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-MLA (Experimental): a fractional 1064-nm neodymium-doped yttrium aluminum garnet (Nd:YAG) picosecond laser with MLA handpiece (P-MLA for short)
  Interventions: Device: a fractional 1064-nm neodymium-doped yttrium aluminum garnet (Nd:YAG) picosecond laser with MLA handpiece
- AF-Er (Sham Comparator): ablative fractional 2940-nm Er:YAG laser (AF-Er for short)
  Interventions: Device: a ablative fractional 2940-nm Er:YAG laser

INTERVENTIONS:
Device: a fractional 1064-nm neodymium-doped yttrium aluminum garnet (Nd:YAG) picosecond laser with MLA handpiece — Picosecond laser is a novel technology characterized by ultra-short, picosecond pulse duration which can be effective for many skin conditions, such as pigmentation, photoaging and wrinkles reduction. When combined with micro-lens array (MLA) optics, high-intensity, micro-injury zones can be generated in the epidermis and dermis, causing optical breakdown of surrounding tissue and stimulating of dermal remodeling with mild side-effects. Previous studies had showed the picosecond lasers with MLA afforded better or similar clinical outcomes as well as fewer side-effects in treating acne scar than non-ablative lasers.
  Arms: P-MLA
Device: a ablative fractional 2940-nm Er:YAG laser — 2940-nm erbium yttrium aluminum garnet (Er:YAG) laser is one of the most commonly used treatments for atrophic acne scars, which can remove the damage tissue of the scars and allow collagen remodeling and re-epithelialization.
  Arms: AF-Er

SUMMARY:
The 1064-nm Nd:YAG picosecond lasers using fractional micro-lens array (P-MLA) was a promising therapy for skin resurfacing. However, no studies have compared P-MLA with ablative fractional 2940-nm Er:YAG lasers (AF-Er) in treating atrophic acne scars. To evaluate the efficacy and safety of P-MLA and AF-Er for the treatment of atrophic acne scars, we performed a prospective, randomized, split-face, controlled trial. Thirty-one Asian patients underwent four consecutive sessions of randomized split-face treatment with P-MLA and AF-Fr at 4-week intervals.

DETAILED DESCRIPTION:
Acne is a common skin disorder affecting 9.38% of the global population, especially among adolescents and young adults. One publication showed that 43% of cases with facial acne could develop scars, and the acne-associated scarring often has a negative effect on patients' psychosocial and physical well-being. A wide range of interventions have been proposed to treat atrophic acne scars, including laser, chemical peels, dermabrasion, injectable fillers and surgical methods. Picosecond laser is a novel technology characterized by ultra-short, picosecond pulse duration which can be effective for many skin conditions, such as pigmentation, photoaging and wrinkles reduction. When combined with micro-lens array (MLA) optics, high-intensity, micro-injury zones can be generated in the epidermis and dermis, causing optical breakdown of surrounding tissue and stimulating of dermal remodeling with mild side-effects. However, there are insufficient prospective comparative studies evaluating the picosecond laser with MLA optics vs. current fractional ablative techniques for the treatment of atrophic acne scars.In this study, we reported a prospective, randomized, split-face, controlled trial that comparing the efficacy and safety of a fractional 1064-nm neodymium-doped yttrium aluminum garnet (Nd:YAG) picosecond laser with MLA handpiece (P-MLA) and ablative fractional 2940-nm Er:YAG laser (AF-Er) for the treatment of atrophic acne scars in Asians.

1. Study design This prospective, randomized, split-face, controlled trial was approved by the Human Ethics Committee of Zhejiang University School of Medicine Second Affiliated Hospital (2022-0419) and performed in accordance with the Declaration of Helsinki. Written informed consent was obtained from all subjects before enrollment.
2. Patient selection A total of thirty-three subjects (16 males and 17 females) aged above 18 years of Fitzpatrick skin types II to type V, with mild to moderate atrophic acne scars were recruited for this study. Inclusion criteria for this study were as follows: (1) age ≥18 years; (2) presence with similar atrophic acne scars on both sides of the face; (3) signed informed consent and cooperated with the follow up and complied the study protocol. Subjects were excluded if they had a previous history of keloid or hypertrophic scar formation, undergone any acne scar treatments in the past 6 months before the first treatment, were pregnant or lactating females, were sensitive to lights, were allergic to lidocaine, had other preexisting skin conditions or uncontrolled systemic diseases.
3. Treatment Enrolled participant was randomized to receive split-face treatment with fractional 1064-nm Nd:YAG picosecond lasers (PicocareTM, Wontech, Korea) on one side and ablative fractional 2940-nm Er:YAG laser (Dermablate MCL31, Asclepion Laser Technologies, Germany) on the other side. The block randomization was used to assign the treatment modality.
4. Assessment Thorough history taking and physical examination were performed in all subjects. Efficacy and safety of the treatments were evaluated at each visit, and VISIA images (Visia CR®; Canfield Scientific, Parsippany, NJ, USA) of front, left and right face were also obtained at both baseline and last visit for final analyses.

Efficacy Efficacy of scar improvement was evaluated by investigators and patients. A blinded investigator assessed the clinical efficacy by the Echelle d'Evaluation Clinique des Cicatrices d'acne (ECCA) grading scale and Investigator's Global Assessment (IGA) scores. ECCA score is calculated on the sum of the number and type of scar (V-type, U-type and M-type)(13). IGA was evaluated using a 5-point scale as follows: 0 = no improvement; 1 = 1-25% improvement; 2 = 26-50% improvement; 3 = 51-75% improvement; 4 = 76-100% improvement. Patients rated their degree of satisfaction about scar improvement, pore, skin texture and overall improvement using a Likert satisfaction scale (1 = very dissatisfied, 2 = dissatisfied, 3 = slightly satisfied, 4 = satisfied, 5 = very satisfied). The primary endpoints were the change of ECCA score, IGA score and degree of patient's satisfaction at the final visit compared the baseline score. We also used VISIA system to evaluate the pore and skin texture objectively.

Safety Patients were evaluated at each session immediately for adverse effects including pain, erythema, edema, exudation, pinpoint bleeding and petechiae. The pain was evaluated using a visual analog scale (VAS) ranging from 0 (no pain) to 10 (unbearable pain). Other immediate adverse effects were recorded with a 0-to-3 severity scale (0 = none; 1 = mild; 2 = moderate; 3 = severe). At next follow-up, patients were also asked to record and document their recovery times and possible long-term adverse effects, including crust shedding time, duration of erythema and edema, post inflammatory hyperpigmentation (PIH), scarring formation, pruritus and milia.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* presence with similar atrophic acne scars on both sides of the face;
* signed informed consent and cooperated with the follow up and complied the study protocol.

Exclusion Criteria:

* a previous history of keloid or hypertrophic scar formation;
* undergone any acne scar treatments in the past 6 months before the first treatment;
* pregnant or lactating females;
* sensitive to lights;
* allergic to lidocaine;
* other preexisting skin conditions or uncontrolled systemic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of scar improvement evaluated by investigators | 8 weeks after final treatment
  the Echelle d'Evaluation Clinique des Cicatrices d'acne (ECCA) grading scale and Investigator's Global Assessment (IGA) scores
Efficacy of scar improvement evaluated by patients | 8 weeks after final treatment
  a Likert satisfaction scale (1 = very dissatisfied, 2 = dissatisfied, 3 = slightly satisfied, 4 = satisfied, 5 = very satisfied)

SECONDARY OUTCOMES:
Adverse effects of pain, erythema, edema, exudation, pinpoint bleeding and petechiae | Immediately after treatment.
  Pain, erythema, edema, exudation, pinpoint bleeding and petechiae
Adverse effects of crust shedding time, duration of erythema and edema, post inflammatory hyperpigmentation (PIH), scarring formation, pruritus and milia. | Through study completion, 8 weeks after final treatment
  crust shedding time, duration of erythema and edema, post inflammatory hyperpigmentation (PIH), scarring formation, pruritus and milia.

CONTACTS AND LOCATIONS:
Overall Officials: Dai Ru, Ph.D, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai R, Cao Y, Su Y, Cai S. Comparison of 1064-nm Nd:YAG picosecond laser using fractional micro-lens array vs. ablative fractional 2940-nm Er:YAG laser for the treatment of atrophic acne scar in Asians: a 20-week prospective, randomized, split-face, controlled pilot study. Front Med (Lausanne). 2023 Nov 16;10:1248831. doi: 10.3389/fmed.2023.1248831. eCollection 2023. PMID 38034535